CLINICAL TRIAL: NCT06225752
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized Clinical Trial of Probucol in Reducing the Risk of Recurrent Stroke in Patients With Symptomatic Intracranial and Extracranial Large-artery Stenosis
Brief Title: Probucol for Symptomatic Intracranial and Extracranial Artery Stenosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023AH040246
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Ischemic Stroke; TIA
Keywords: Probucol; Recurrent stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Probucol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probucol Group (Experimental): The study drug should be started as soon as possible within 7 days after symptom onset.
  Interventions: Drug: Probucol
- Placebo Probucol Group (Placebo Comparator): The study drug should be started as soon as possible within 7 days after symptom onset.
  Interventions: Drug: Placebo probucol

INTERVENTIONS:
Drug: Probucol — Inclusion Days 1-30: Probucol 1000mg/day (500mg per dose, twice daily, a minimum of 4 hours should elapse between each pair of doses.) Inclusion Days 31 and beyond: Probucol 500mg/day (250mg per dose, twice daily, a minimum of 4 hours should elapse between each pair of doses.)
  Arms: Probucol Group
Drug: Placebo probucol — Inclusion Days 1-30: Placebo Probucol 1000mg/day (500mg per dose, twice daily, a minimum of 4 hours should elapse between each pair of doses.) Inclusion Days 31 and beyond: Placebo Probucol 500mg/day (250mg per dose, twice daily, a minimum of 4 hours should elapse between each pair of doses.)
  Arms: Placebo Probucol Group

SUMMARY:
This study is a multicenter, double-blind, placebo-controlled, randomized clinical trial that aims to evaluate the efficacy of probucol on the reduction of the risk of recurrent stroke in patients with symptomatic intracranial or extracranial arterial stenosis.

DETAILED DESCRIPTION:
This study is a multicenter, double-blind, placebo-controlled, randomized clinical trial that aims to evaluate the efficacy of probucol on the reduction of the risk of recurrent stroke in patients with symptomatic intracranial or extracranial arterial stenosis. During the study period, 5452 patients at intermediate risk for ischemic stroke or TIA will be enrolled from 100 centers.To evaluate whether probucol, as compared with placebo, reduces the risk of recurrent stroke in patients at high risk for ischemic stroke or TIA within 7 days of onset.Patients in one arm will receive probucol initiated with a dose of 1000 mg per day on days 1 through 30, and continuing with 500 mg per day after day 31, and those in the other arm will receive an equivalent placebo drug. Study visits will be performed on the day of randomization, at discharge, at day 90 and at 1 year and then followed up annually until the occurrence of the endpoint event or the end of the study. In addition, patients will be followed up at any time when new clinical symptoms of the neurologic system and suspicious events occur, including worsening of the original ischemic event and the appearance of new transient or persistent neurologic symptoms.

ELIGIBILITY:
Inclusion Criteria:

1.40 years or older than 40 years; 2.Ischemic stroke or transient ischemic attack (TIA); 3.Within 7 days from onset to randomization; 4.Main intracranial or extracranial arteries supplying the ischemic event region are narrowed by more than 50%; 5.Informed consent signed.

Exclusion Criteria:

1. Presumed cardiac source of embolus, such as atrial fibrillation, prosthetic cardiac valve, endocarditis or patent foramen ovale;
2. Stroke/TIA due to arterial dissection, angioplasty, or vascular surgery;
3. Usage of probucol within 30 days before randomization;
4. Known allergy or sensitivity or intolerance to probucol;
5. Myocardial disease within the past 30 days, including myocardial infarction, myocarditis;
6. With ventricular tachycardia, bradycardia, tip-twist ventricular tachycardia；
7. With Q-Tc interval prolongation, or currently using drugs that may cause Q-Tc interval prolongation (male Q-Tc>450ms, female Q-Tc>470ms);
8. Cardiac syncope or unexplained syncope;
9. Impaired hepatic (ALT or AST > twice the upper limit of normal range) or kidney (creatinine exceeding 1.5 times of the upper limit of normal range or eGFR less than 50 ml/min) function at randomization;
10. Anemia (haemoglobin <10g/dL), thrombocytopenia (platelet count <100×109/L) or leucopenia (white blood cell <3×109/L) at randomization;
11. Planned surgery or interventional treatment requiring cessation of the study drug during the study;
12. Participating in another clinical trial with an investigational drug or device concurrently or during the last 30 days;
13. Pregnant or lactating women; Pregnant, currently trying to become pregnant, or of child-bearing potential and not using birth control;
14. Severe non-cardiovascular comorbidity with a life expectancy of less than 1 years;
15. Serious drug or alcohol abuse in the past 1 year；
16. Inability to understand and/or follow research procedures due to mental, cognitive, or emotional disorders, or to be an unsuitable candidate for the study for any other considered by the investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5452 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Recurrent stroke event | within 1 year
  Ischemic or hemorrhagic stroke

SECONDARY OUTCOMES:
Recurrent ischemic stroke event | within 1 year
  Incidence of any new ischemic stroke
Composite vascular events | within 1 year
  Including ischemic stroke, hemorrhagic stroke, myocardial infarction and vascular death
Poor functional outcome | within 1 year
  Defined as a modified Rankin Scale (mRS) score ≥3(The mRS Scale is used to evaluate the recovery of neurological function in stroke patients. It consists of a seven-point scale, with Grade 0 indicating no symptoms at all. Grade 1 represents the presence of symptoms but without significant disability, allowing for the performance of regular jobs and activities. Grade 2 signifies mild disability where individuals are unable to perform all work and activities but can manage personal affairs independently. Grade 3 indicates moderate disability requiring assistance from others for walking without aid. Grade 4 denotes severe disability where individuals cannot walk unassisted and are unable to care for their own needs. Grade 5 represents severe disability with bedridden status, incontinence, and necessitating continuous care round-the-clock. Finally, Grade 6 signifies death.)
All-cause mortality | within 1 year
  Death from any cause

OTHER OUTCOMES:
Change in levels of oxidized low-density lipoprotein cholesterol (Ox-LDL) | within 1 year
  Ox-LDL is a component specific to the atherosclerotic lesion area that is not present in normal arterial vascular tissue and is elevated in atherosclerotic strokes
Change in the rate of responsible vessel stenosis | within 1 year
  Stenosis of the responsible vessel at enrollment >50%
Adverse events | within 1 year
  The difference in the proportion of adverse events (AEs) between Probucol and the placebo group
Severe adverse events | within 1 year
  The difference in the proportion of serious adverse events (SAEs) between Probucol and the placebo group;

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affliated Hospital of Wannan Medical College, Wuhu, China

IPD SHARING:
Plan to Share IPD: No